CLINICAL TRIAL: NCT00766155
Title: Preoperative Chemoradiotherapy and Postoperative Chemotherapy With Capecitabine and Oxaplatin vs.Capecitabine Alone in Locally Advanced Rectal Cancer (PETACC-6)
Brief Title: Chemotherapy and Radiation Therapy Before Surgery Followed by Capecitabine With or Without Oxaliplatin in Treating Patients With Locally Advanced Rectal Cancer
Acronym: PETACC-6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-40054-22062; EU-20880; PETACC-6; ROCHE-EORTC-40054; 2006-006532-21 (EudraCT Number)
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin

ARMS (2):
- Arm I (Active Comparator): Patients receive oral capecitabine twice daily and undergo concurrent 3-dimensional conformal radiotherapy 5 days a week on days 1-33. Patients may receive additional chemoradiotherapy on days 36-38. Patients then undergo surgery. Beginning 4-8 weeks after surgery, patients receive capecitabine twice daily on day 1-15. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: capecitabine
- Arm II (Experimental): Patients receive oral capecitabine twice daily and undergo concurrent 3-dimensional conformal radiotherapy 5 days a week on days 1-33. Patients also receive oxaliplatin IV over 1 hour on days 1, 8, 15, 22, and 29 prior to radiotherapy followed by surgery. Patients may receive additional chemoradiotherapy on days 36-38. Beginning 4-8 weeks later, patients receive oxaliplatin IV over 2 hours on day 1, and oral capecitabine twice daily on days 1-15. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: capecitabine; Drug: oxaliplatin

INTERVENTIONS:
Drug: capecitabine — Given orally
Drug: oxaliplatin — Given IV
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy that uses a 3-dimensional image of the tumor to help focus thin beams of radiation directly on the tumor may kill more tumor cells and have fewer side effects. Giving chemotherapy together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether capecitabine is more effective with or without oxaliplatin in treating patients with rectal cancer.

PURPOSE: This randomized phase III trial is studying giving chemotherapy together with radiation therapy before surgery followed by capecitabine with or without oxaliplatin to see how well it works in treating patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Investigate whether the addition of oxaliplatin to neoadjuvant chemoradiotherapy and adjuvant chemotherapy comprising capecitabine improves disease-free survival in patients with locally advanced rectal cancer.

Secondary

* Compare the overall survival of patients with locally advanced rectal cancer treated with neoadjuvant chemoradiotherapy and adjuvant chemotherapy comprising capecitabine with versus without oxaliplatin.
* Determine the loco-regional failure and distant failure of patients treated with these regimens.
* Determine the pathological down-staging (ypT0-2N0) of patients treated with these regimens.
* Determine the pathological complete remission (yp T0N0) rate of patients treated with these regimens.
* Determine the tumor progression grade and histopathological R0 resection of patients treated with these regimens.
* Determine the sphincter preservation rate of patients treated with these regimens.
* Determine the perioperative complication rate of these regimens in these patients.
* Determine the toxicity of these regimens in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to treating center, clinical T category (T1-3 vs T4), clinical nodal status (Nx vs NO vs N1-2), distance from the tumor to the anal verge (≤ 5 cm vs > 5 cm) and method of locoregional staging (EUS+MRI vs EUS+CTscan vs MRI alone). Patients are randomized to 1 of 2 treatment arms.

* Arm I (control):

  * Neoadjuvant therapy: Patients receive oral capecitabine twice daily on days 1-35. Patients also undergo concurrent 3-dimensional conformal radiotherapy 5 days a week on days 1-33 followed by surgery. Patients may receive additional chemoradiotherapy on days 36-38.
  * Adjuvant therapy: Beginning 4-8 weeks after surgery, patients receive oral capecitabine twice daily on days 1-15. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (investigational):

  * Neoadjuvant therapy: Patients receive oral capecitabine twice daily and undergo concurrent 3-dimensional conformal radiotherapy 5 days a week on days 1-33. Patients also receive oxaliplatin IV over 1 hour on days 1, 8, 15, 22, and 29 prior to radiotherapy followed by surgery. Patients may receive additional chemoradiotherapy on days 36-38.
  * Adjuvant therapy: Beginning 4-8 weeks after surgery, patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-15. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months for 3 years, and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum

  * Tumor ≤ 12 cm from the anal verge
  * Stage T3-4 or any node-positive disease
* No evidence of metastatic disease (confirmed by negative CT scan of the chest and abdomen)
* Resectable disease or expected to become resectable after preoperative chemoradiation
* May only be randomized once in this trial

PATIENT CHARACTERISTICS:

* WHO/ECOG performance status 0-2
* Hemoglobin ≥ 10.0 g/dL (transfusion allowed to achieve or maintain levels)
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* ALT and AST ≤ 2.5 times upper level of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Total bilirubin ≤ 1.5 times ULN
* Creatinine clearance > 50 mL/min
* Creatinine ≤ 1.5 times ULN
* Able to swallow tablets
* No prior or concurrent malignancies within the past 5 years except for adequately treated cone-biopsied carcinoma in situ of the cervix or basal cell carcinoma of the skin
* No clinically significant (i.e., active) cardiac disease, including any of the following:

  * Congestive heart failure
  * Symptomatic coronary artery disease
  * Cardiac arrhythmia
* No myocardial infarction within the past 12 months
* No known significant impairment of intestinal resorption (e.g., chronic diarrhea, inflammatory bowel disease)
* No pre-existing conditions that would preclude chemoradiotherapy or radiotherapy (i.e., fistulas, severe ulcerative colitis [particularly patients currently taking sulfasalazine], Crohn's disease, or prior adhesions)
* No peripheral neuropathy ≥ grade 2 by CTCAE v3.0
* No serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease
* No history of uncontrolled seizures, central nervous system disorders or psychiatric disability that, in the opinion of the principal investigator, is clinically significant and would preclude giving informed consent or interfere with compliance with oral drug administration
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior cytotoxic chemotherapy or radiation therapy for rectal cancer
* No prior radiation therapy to the pelvis
* No prior or concurrent investigational drug, agent, or procedure
* More than 4 weeks since prior participation in the active or follow-up period of another investigational protocol
* No known allergy or any other adverse reaction to any of the study drugs or to any related compound
* No known dihydropyrimidine dehydrogenase deficiency
* No organ allograft requiring immunosuppressive therapy
* No concurrent sorivudine or chemically related analogues (e.g., brivudine)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1094 (Actual)
Dates: Start 2008-08; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Overall survival within at least the first 5 years after treatment
Loco-regional failure, defined as local or regional recurrence, inoperable disease, or R1 or R2 resection
Distant failure (i.e., distant metastasis)
Pathological down-stage (ypT0, 2N0) rate
Pathological complete remission (ypT0N0) rate
Tumor regression grade
Histopathological R0 resection rate
Sphincter preservation rate
Preoperative complication rate
Toxicity according to CTCAE v.3.0 weekly during treatment, at 4-8 weeks after surgery, at therapy completion, and every 6 months for 5 years after therapy completion

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joachim Schmoll, MD, PhD, Study Chair — Martin-Luther-Universität Halle-Wittenberg; Karin Haustermans, Study Chair — U.Z. Gasthuisberg, Leuven

REFERENCES:
- [Derived] Schmoll HJ, Stein A, Van Cutsem E, Price T, Hofheinz RD, Nordlinger B, Daisne JF, Janssens J, Brenner B, Reinel H, Hollerbach S, Caca K, Fauth F, Hannig CV, Zalcberg J, Tebbutt N, Mauer ME, Marreaud S, Lutz MP, Haustermans K. Pre- and Postoperative Capecitabine Without or With Oxaliplatin in Locally Advanced Rectal Cancer: PETACC 6 Trial by EORTC GITCG and ROG, AIO, AGITG, BGDO, and FFCD. J Clin Oncol. 2021 Jan 1;39(1):17-29. doi: 10.1200/JCO.20.01740. Epub 2020 Oct 1. PMID 33001764